CLINICAL TRIAL: NCT06739538
Title: Effects Of Bobath Exercises Combined With Gasotransmitter On Spastic Diplegic CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/752
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Gasotransmitters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath exercises (Experimental)
  Interventions: Diagnostic Test: Bobath exercises
- Gasotransmitters (Active Comparator)
  Interventions: Combination Product: Gasotransmitters

INTERVENTIONS:
Diagnostic Test: Bobath exercises — Bobath concept, are therapeutic techniques designed to improve motor control and function in individuals with neurological conditions, particularly those with cerebral palsy. These exercises focus on facilitating normal movement patterns, enhancing postural stability, and reducing muscle spasticity. The approach emphasizes individualized treatment, utilizing hands-on techniques to promote movement awareness and encourage the development of functional skills. By reinforcing weak movements and inhibiting overactive ones, Bobath exercises aim to enhance overall motor abilities and improve the quality of life for affected individuals.
  Arms: Bobath exercises
Combination Product: Gasotransmitters — such as nitric oxide (NO), carbon monoxide (CO), and hydrogen sulfide (H₂S), are small gaseous signaling molecules that play key roles in various physiological functions, including the regulation of muscle tone and neuroinflammation. In the context of spastic diplegic cerebral palsy (CP), gasotransmitters may help reduce spasticity and pain. Gasotransmitters help reduce spasticity and pain in children with spastic diplegic cerebral palsy through multiple mechanisms: Muscle relaxation and improved blood flow reduce muscle tightness, Anti-inflammatory and neuroprotective properties help minimize the damage that exacerbates spasticity.They also modulate pain pathways, both centrally and peripherally, reducing pain perception.
  Arms: Gasotransmitters

SUMMARY:
This study examines the effects of combining Bo bath neurodevelopmental exercises with gasotransmitter in children with spastic diplegic cerebral palsy, a condition marked by muscle stiffness and coordination challenges in the legs.

DETAILED DESCRIPTION:
The primary objective is to enhance motor learning by reinforcing weak movement patterns while reducing excessive muscle activity. Additionally, this combination aims to improve postural control, movement coordination, and overall functional abilities.The randomized controlled trial includes 47 children aged 6-18, divided into three groups: one receiving only Bo bath exercises, another receiving gasotransmitter alone, and a third receiving both interventions. Baseline assessments were conducted, and ethical approval along with informed consent was obtained. The interventions target spasticity reduction and gross motor improvement, with outcomes measured using the Gross Motor Function Classification System (GMFCS) for motor skills and the Modified Ashworth Scale for spasticity. Findings suggest that combining Bo bath therapy with gasotransmitters effectively reduces spasticity, enhances motor control, and supports activities of daily living, highlighting its potential as an effective therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* A Confirmed diagnosis of spastic diplegic cerebral palsy
* Participants aged 6 to 18 years.
* Moderate to severe spasticity in the lower limbs, as measured by the Modified Ashworth Scale.
* Ability to follow simple instructions and participate in the stretching exercises.
* Written informed consent obtained from the participant's legal guardian or the participant if of legal consenting age.
* No significant changes in medication or therapy for cerebral palsy in the three months prior to the study.

Exclusion Criteria:

* Presence of other neurological conditions apart from spastic diplegic cerebral palsy.
* History of major orthopaedic surgery in the past year or planned surgery during the study period.
* Receipt of botulinum toxin injections in the lower limbs within the last six months.
* Severe joint contractures that limit the range of motion necessary for the stretching exercises.
* Any medical condition that contraindicates participation in the study, such as uncontrolled epilepsy, severe cardiovascular disorders, or acute infections.
* Inability or unwillingness to comply with the study protocol and scheduled visits.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | 12 Months
  The Gross Motor Function Classification System (GMFCS) is a five-level clinical classification tool that categorizes the gross motor function of children and young people with cerebral palsy (CP) based on their self-initiated movement abilities, particularly sitting, walking, and mobility. The GMFCS is used to understand and predict the mobility needs and functional capabilities of individuals, aiding in treatment planning, goal setting, and tracking functional changes over time.
Manual Muscle Testing Manual Muscle Testing (MMT) | 12 months
  It is a clinical assessment technique used to evaluate and grade the strength of individual muscles or muscle groups based on their ability to resist force. In MMT, the clinician applies pressure to a muscle while the patient resists, allowing for a standardized rating, typically on a scale from 0 to 5:

CONTACTS AND LOCATIONS:
Locations (1):
- Ilaj Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No